CLINICAL TRIAL: NCT01020188
Title: A Pilot Study Investigating the Role of Thrombin Generation and Rotational Thromboelastometry in Assessing the Prothrombotic Phenotype of Paroxysmal Nocturnal Haemaglobinuria
Brief Title: Study of Global Coagulation Tests in Patients With Paroxysmal Nocturnal Haemoglobinuria
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Dr Raj Patel, King's College Hospital NHS Foundation Trust
Other Study IDs: KCH1125
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Paroxysmal Nocturnal Haemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Paroxysmal nocturnal haemaoglobinuria (PNH) is a rare disease which results in breakdown of the red blood cells and bone marrow failure. It is associated with an increased risk of blood clots. Until recently, treatment has been with blood transfusions and in patients with a blood clot, blood thinners. A new treatment called eculizumab is now standard for patients who require regular blood transfusions. It works in the majority of patients by preventing the breakdown of red blood cells. This can eliminate the need for blood transfusion and reduce the risk of blood clots. It is not well understood why patients with PNH are at high risk of blood clots. The investigators plan to use specialised blood tests to assess the stickiness of the blood before starting eculizumab treatment and monthly after starting treatment. The investigators will compare these tests with standard tests of clotting.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a PNH clone

Exclusion Criteria:

* Longterm anticoagulation for previous venous thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with paroxysmal nocturnal haemoglobinuria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To establish the role of thrombin generation in assessing the prothrombotic phenotype of PNH | After sample is obtained

SECONDARY OUTCOMES:
To establish the role of thromboelastometry in evaluating the prothrombotic phenotype of PNH | After sample is obtained
To establish effects of eculizumab treatment on thrombin generation and thromboelastometry | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raj K Patel, MD, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Trust, London, United Kingdom